CLINICAL TRIAL: NCT00835328
Title: Role of Glucagon-Like Peptide-1 (GLP-1) in Congenital Hyperinsulinism: Effect of Exendin (9-39) on Glucose Requirements to Maintain Euglycemia
Brief Title: Effect of Exendin (9-39) on Glucose Requirements to Maintain Euglycemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped prematurely to test a new formulation of Exendin (9-39)
Sponsor: Diva De Leon (Other)
Responsible Party: Sponsor-Investigator, Diva De Leon, Professor of Pediatrics, Children's Hospital of Philadelphia, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008-10-6256
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Congenital Hyperinsulinism
Keywords: Congenital Hyperinsulinism; Hyperinsulinism; Hypoglycemia; KATP channel; Metabolic Diseases; Pancreatic Disease; Glucose Metabolism Disorders; Infant, Newborn, Diseases
MeSH Terms: conditions — Congenital Hyperinsulinism; Hyperinsulinism; Hypoglycemia; Metabolic Diseases; Pancreatic Diseases; Glucose Metabolism Disorders; Infant, Newborn, Diseases | interventions — exendin (9-39)

STUDY DESIGN:
Intervention Model Description: This is a two-period, two-treatment cross-over clinical study with a dose-escalation component. Each subject, in random order, will receive an intravenous (IV) infusion of Exendin (9-39) and normal saline vehicle for up to 9 hours on two separate days.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exendin (9-39) 0.02 mg/kg/hr (Experimental): Cohort 1: Participants will be administered 0.02 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 9 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first). Glucose infusion rates (GIR) will be titrated three hours prior to infusions to keep blood glucose in the range of 70-90 mg/dL. During both infusions, blood glucose will be measured every 30 minutes.
  Interventions: Drug: Exendin (9-39); Drug: Vehicle
- Exendin (9-39) 0.04 mg/kg/hr (Experimental): Cohort 2: Participants will be administered 0.04 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 9 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first). Glucose infusion rates (GIR) will be titrated three hours prior to infusions to keep blood glucose in the range of 70-90 mg/dL. During both infusions, blood glucose will be measured every 30 minutes.
  Interventions: Drug: Exendin (9-39); Drug: Vehicle
- Exendin (9-39) 0.10 mg/kg/hr (Experimental): Cohort 3: Participants will be administered 0.10 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 6 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first). Glucose infusion rates (GIR) will be titrated three hours prior to infusions to keep blood glucose in the range of 70-90 mg/dL. During both infusions, blood glucose will be measured every 30 minutes.
  Interventions: Drug: Exendin (9-39); Drug: Vehicle
- Exendin (9-39) 0.20 mg/kg/hr (Experimental): Cohort 4: Participants will be administered 0.20 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 9 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first). Glucose infusion rates (GIR) will be titrated three hours prior to infusions to keep blood glucose in the range of 70-90 mg/dL. During both infusions, blood glucose will be measured every 30 minutes.
  Interventions: Drug: Exendin (9-39); Drug: Vehicle

INTERVENTIONS:
Drug: Exendin (9-39) — A short-term intravenous infusion of the investigational drug, Exendin (9-39), will be administered over up to 9 hours.
Drug: Vehicle — A short-term intravenous infusion of normal saline (0.9% NaCl), or the vehicle, will be administered over up to 9 hours.
  Other Names: Placebo

SUMMARY:
The primary aim of this study is to evaluate the effect of Exendin (9-39) on glucose requirements to maintain euglycemia in pediatric patients with congenital hyperinsulinism (CHI) who have failed medical therapy. The secondary aims are to determine the therapeutic plasma levels, plasma half-life and pharmacokinetics of Exendin (9-39) during a 9-hour intravenous infusion.

DETAILED DESCRIPTION:
This study will enroll infants with congenital hyperinsulinism owing to KATP channel mutations who are unresponsive to medical therapy and will require a pancreatectomy to control hypoglycemia from a single academic medical center in the United States.

An open-label, two-period, two-treatment crossover study design with a dose-escalation component will be implemented. Successive cohorts of patients (up to 5 participants/cohort) will each receive a fixed dose of Exendin (9-39) infusion and normal saline vehicle on two separate days in random order. The protocol specifies 0.02 mg/kg/hr, via continuous intravenous infusion, administered over 9-hours for the first cohort. The volume of saline to be infused will be calculated to match the volume of Exendin (9-39). Successive cohorts will be given doses that are increased in up to 1/2 log increments. Overall, the investigators hypothesize that antagonism of the GLP-1 receptor by Exendin (9-39) will increase fasting blood glucose levels, prevent protein-induced hypoglycemia and decrease glucose requirement to maintain euglycemia in infants with CHI.

Aim 1. To examine the effect of Exendin (9-39) on glucose requirements to maintain euglycemia in infants with congenital hyperinsulinism unresponsive to medical therapy.

Aim 2. To determine therapeutic plasma levels, plasma half-life and pharmacokinetics of Exendin-(9-39) during an intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed clinical diagnosis of congenital hyperinsulinism
2. Infants less than 12 months of age at study enrollment
3. Failure to respond to treatment with diazoxide

Exclusion Criteria:

1. Evidence of a medical condition that might alter results, including kidney failure, severe liver dysfunction, severe respiratory or cardiac failure
2. Treatment with medications that may affect glucose metabolism at the time of initiation of study procedures, including:

   1. Treatment with glucagon 4 hours prior to infusion (T=0)
   2. Treatment with octreotide 24 hours prior to infusion (T=0)
   3. Treatment with diazoxide 72 hours prior to infusion (T=0)
3. Suspected Beckwith-Wiedemann syndrome or other syndromic forms of congenital hyperinsulinism.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2009-08-26 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diva D De Leon, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on a confirmed clinical diagnosis of congenital hyperinsulinism at 1 academic medical center between August 2009 and October 2019. The first participant was enrolled on August 26, 2008 and the last participant was enrolled in January 25, 2017.
Pre-assignment Details: Of the 14 enrolled participants, 13 met inclusion criteria and were randomized to treatment.
Period: Cohort 1: Dose Level 1
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr
Started | 5 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 2
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr
Started | 0 | 2 | 0 | 0
Completed | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3: Dose Level 3
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr
Started | 0 | 0 | 2 | 0
Completed | 0 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 4: Dose Level 4
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr
Started | 0 (Cohort#4 enrolled 4 subsequent subjects) | 0 | 0 | 4
Completed | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exendin (9-39) 0.02 mg/kg/hr: Cohort 1: Participants will be administered 0.02 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 9 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first).
- Exendin (9-39) 0.04 mg/kg/hr: Cohort 2: Participants will be administered 0.04 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 9 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first).
- Exendin (9-39) 0.10 mg/kg/hr: Cohort 3: Participants will be administered 0.10 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 6 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first).
- Exendin (9-39) 0.20 mg/kg/hr: Cohort 4: Participants will be administered 0.20 mg/kg/hr of Exendin (9-39) and vehicle (normal saline), via continuous intravenous infusion, over 9 hours on two separate days in random order, with 3 hours of follow-up after the last dose is administered or until blood glucose is < 70 mg/dL (whichever comes first).
- Total: Total of all reporting groups
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Total
Number analyzed (Participants) | 5 | 2 | 2 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 2 | 2 | 4 | 13
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 1 | 7
  Male | 1 | 1 | 1 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 4 | 2 | 2 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 2 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 01 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Glucose Infusion Rate (GIR)
Description: To assess the effect of Exendin (9-39) on glucose infusion rate, glucose infusion rate (GIR) over the last 2 hours of the treatment period was calculated by adding the total amount of intravenous glucose (mg) received over 2 hours divided by the weight (kg) and by time (120 min) during infusion of Exendin (9-39) and normal saline vehicle.
Time Frame: Up to 9 hours after the initiation of infusion
Population: Subjects served as their own control for comparison between the effects of Exendin (9-39) and the normal saline vehicle. The trial was terminated after 14 participants enrolled in the study. No data is available for any outcome measures.
Groups:
- Vehicle: All participants will be administered normal saline vehicle, via continuous intravenous infusion, over up to 9 hours. Subjects served as their own control for comparison between the effects of Exendin (9-39) and the normal saline vehicle.
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: To Determine the Pharmacokinetics of Exendin (9-39)
Description: The following PK variables of interest include AUC0-∞, AUC0-t, maximal concentration (Cmax), time to maximal concentration (Tmax), concentration at end of infusion (Ceoi), steady state volume of distribution (Vss), clearance (CL) and half-life (t1/2) of Exendin (9-39). These will be derived through both non-compartmental and model-based methods.
Time Frame: Up to 12 hours after the initiation of infusion
Population: as for outcome 1
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Safety and Tolerability of Exendin (9-39)
Description: Number of participants with adverse events as a measure of safety and tolerability [evaluated by the result of laboratory safety tests (hematology, chemistry, urinalysis), vital signs, physical examinations, and 12-lead ECG]
Time Frame: Up to 24 hours post-infusion
Population: as for outcome 1
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Mean Plasma Insulin
Description: To assess the effect of Exendin (9-39) on plasma insulin levels, samples were collected at various time points during the infusion [Exendin (9-39) or vehicle] including: at the start of the infusion (T=0) and at 1, 5, and 9 hours post initiation of the infusion.
Time Frame: Up to 9 hours after the initiation of infusion
Population: as for outcome 1
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Plasma Glucose
Description: To assess the effect of Exendin (9-39) on plasma glucose levels, samples were collected at various time points during the infusion [Exendin (9-39) or vehicle] including: at the start of the infusion (T=0) and at 1, 5, and 9 hours post initiation of the infusion.
Time Frame: Up to 9 hours after the initiation of infusion
Population: as for outcome 1
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Mean Betahydroxybutyrate Levels
Description: To assess the effect of Exendin (9-39) on mean betahydroxybutyrate levels, samples were collected at various time points during the infusion [Exendin (9-39) or vehicle] including: at the start of the infusion (T=0) and hourly up to 12-hours post initiation of the infusion.
Time Frame: Up to 12 hours after the initiation of infusion
Population: as for outcome 1
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety monitoring for adverse events will occur for 24-hours post study-drug infusion. For this study, the treatment follow-up period is defined by the half-life of the investigational product.
Description: Safety population = all participants who received any dose of the investigational product. Subjects served as their own control for comparison between the effects of Exendin (9-39) and the normal saline vehicle.
Groups:
- Vehicle: All participants will be administered normal saline vehicle via continuous intravenous infusion.
Arm/Group | Exendin (9-39) 0.02 mg/kg/hr | Exendin (9-39) 0.04 mg/kg/hr | Exendin (9-39) 0.10 mg/kg/hr | Exendin (9-39) 0.20 mg/kg/hr | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/2 | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/2 | 0/4 | 0/13
Other Adverse Events (participants affected / at risk) | 1/5 | 2/2 | 2/2 | 4/4 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exendin (9-39) 0.02 mg/kg/hr (N=5) | Exendin (9-39) 0.04 mg/kg/hr (N=2) | Exendin (9-39) 0.10 mg/kg/hr (N=2) | Exendin (9-39) 0.20 mg/kg/hr (N=4) | Vehicle (N=13)
Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 8 (8)
Abormal Lab Value - AST (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated after 14 participants enrolled in the study. No data is available for any outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT00835328/Prot_SAP_000.pdf